CLINICAL TRIAL: NCT03015363
Title: Comparison, Calibration, and Validation of the Non-invasive Cloud DX Pulsewave Health MonitorTM With Direct Invasive Radial and Central Arterial Measurements During Cardiac Catheterization
Brief Title: Clinical Calibration & Validation of a Next-Generation Blood Pressure Monitor for Patient Management
Acronym: CCV
Status: Completed | Type: Observational
Sponsor: Cardiovascular Research New Brunswick (Other)
Collaborators: Horizon Health Network (Other); Dalhousie University (Other); Cloud DX Inc. (Industry); New Brunswick Health Research Foundation (Other)
Responsible Party: Principal Investigator, Sohrab Lutchmedial, MD, FRCPC, Co-Director of CVR-NB/ Director of NBHC Catheterization Laboratory, Cardiovascular Research New Brunswick
Other Study IDs: RS#: 2013-1919
Record Dates: First submitted 2017-01-05; First posted 2017-01-10 (Estimated); Results first posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Hypertension
Keywords: Hypertension; Telemonitoring; Vital signs
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the Cloud DX Pulsewave Health Monitor study is to prospectively calibrate and validate a novel, non-invasive wrist cuff blood pressure device against the gold standard for hemodynamic monitoring (intra-arterial pressure) in voluntarily consented patient participants who are scheduled for an elective cardiac catheterization procedure for clinically valid reasons.

DETAILED DESCRIPTION:
The Cloud DX Pulsewave Health Monitor is a non-invasive wrist cuff blood pressure device that is licensed by Health Canada with Food and Drug Administration approval. Systolic and diastolic pressures are measured via the arterial pulse waveform of the left radial artery. Initially, the blood pressure algorithm was created and calibrated using the auscultatory method. The purpose of this study is to calibrate the device to the clinical gold standard of peripheral and central intra-arterial pressures.

The device acquires a pulse signal in real-time, stores signal and measurement data, and displays stored signal and measurement data for interpretation via internet servers where it is accessible by end-users (physicians and/or patients). The system provides secure accounts for both in-patient and out-patient monitoring. Cloud DX's Pulsewave Health Monitor servers are housed in a secure data center. Privacy measures are to SSAE16 SOC-1 Type-II compliance: 1) restricted secure access, 2) dedicated firewall, 3) HTTPS channel communication via website, 4) self-encrypting hard-drives rendered useless if removed from the server.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 19 years of age
* Patients recommended by their cardiologist for a first-time, elective cardiac catheterization procedure
* Wrist circumference between 13.5cm - 23cm (5.3 - 9.1in.)
* Bilateral arm blood pressure equality (systolic within ±10mmHg; diastolic within ±5mmHg) on 2 separate readings (Nurse Associate & TRA)
* Willing to volunteer to participate and to sign the study specific informed consent form

Exclusion Criteria:

* No history of peripheral vascular disease, no previous percutaneous coronary intervention, nor previous coronary artery bypass graft
* No arrhythmia
* No abdominal aortic aneurysm
* No hand/body tremor

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for an elective, non-emergent cardiac catheterization with right radial access; exclusion criteria being no history of peripheral vascular disease, no previous coronary artery bypass graft, no precious percutaneous coronary intervention, abdominal aortic aneurysm, arrhythmia, hand/body tremor, nor bilateral arm pressure inequality during history and physical.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sohrab Lutchmedial, MD, FRCPC, Principal Investigator — Cardiovascular Research New Brunswick
Locations (1):
- Horizon Health Network, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Melville S, Teskey R, Philip S, Simpson JA, Lutchmedial S, Brunt KR. A Comparison and Calibration of a Wrist-Worn Blood Pressure Monitor for Patient Management: Assessing the Reliability of Innovative Blood Pressure Devices. J Med Internet Res. 2018 Apr 25;20(4):e111. doi: 10.2196/jmir.8009. PMID 29695375
- See also: Device company website — http://www.clouddx.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 37 eligible patients voluntarily consented to participate in the study, although 3 participants withdrew and 14 participants failed to meet the study eligibility criteria.
Groups:
- Prospective Cohort (1): Voluntarily consented patient participants scheduled for an elective, non-emergent cardiac catheterization with right radial access.
Period: Overall Study
Arm/Group | Prospective Cohort (1)
Started | 37
Completed | 20
Not Completed | 17
Not completed — Physician Decision | 14
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Prospective Cohort (1)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 20
Smoking (%) [Count of Participants; unit: Participants] | 3
Diabetes (%) [Count of Participants; unit: Participants] | 7
Dyslipidemia (%) [Count of Participants; unit: Participants] | 14
Hypertension (%) [Count of Participants; unit: Participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: Systolic Pressure
Description: Central aortic pressure (mmHg)
Time Frame: Simultaneous non-invasive blood pressure device and intra-arterial fluid-filled pressure catheter measurements on day of cardiac catheterization procedure.
Population: Voluntarily consented patient participants scheduled for an elective, non-emergent cardiac catheterization with right radial access.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prospective Cohort (1)
Number analyzed (Participants) | 20
mmHg | 133.4 (22.0)

2. Primary Outcome: Diastolic Pressure
Description: Central aortic pressure (mm Hg)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prospective Cohort (1)
Number analyzed (Participants) | 20
mmHg | 67.4 (8.7)

3. Primary Outcome: Systolic Pressure
Description: Peripheral arterial pressure (mm Hg)
Time Frame: Non-invasive blood pressure device measurements on day of cardiac catheterization procedure.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prospective Cohort (1)
Number analyzed (Participants) | 20
mmHg | 145.7 (20.2)

4. Primary Outcome: Diastolic Pressure
Description: Peripheral arterial pressure (mm Hg)
Time Frame: Non-invasive blood pressure device measurements on day of cardiac catheterization procedure.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prospective Cohort (1)
Number analyzed (Participants) | 20
mmHg | 66.2 (9.1)

ADVERSE EVENTS:
Arm/Group | Prospective Cohort (1)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This study was an iterative process in the calibration and validation of the Cloud DX, Inc. Pulsewave Health Monitor oscillometric (automatic) wrist cuff device. The device has not yet been calibrated and validated via the ISO 81060-2_2020 'universal' protocol, although this requirement is currently in progress.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No